CLINICAL TRIAL: NCT01416636
Title: A Double Blind Controlled Clinical Study to Investigate the Efficacy and Tolerability of Subcutaneous Treprostinil Sodium in Patients With Severe Non-operable Chronic Thromboembolic Pulmonary Hypertension (CTREPH)
Brief Title: Efficacy and Tolerability of Subcutaneously Administered Treprostinil Sodium in Patients With Severe (Non-operable) Chronic Thromboembolic Pulmonary Hypertension (CTREPH)
Acronym: CTREPH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SciPharm SàRL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116-02
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Non-operable Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treprostinil sodium low dose - Arm I (Active Comparator): Arm I (low dose):
  Subject was treated with a low dose of Treprostinil sodium. Dose was escalated to an approximate target dose of 3 ng/kg/min after the first 12 weeks and was kept stable for another 12 weeks.
  Due to the predefined infusion rate setting schedule an interim dose of up to 6 ng/kg/min could be reached for few days at the end of the phases 1,2 and 3.
  This depended on the patient's exact weight and is caused by the limited infusion rate setting possibility of the infusion pump.
  Interventions: Drug: Treprostinil sodium
- Treprostinil sodium high dose - Arm II (Experimental): Subject was treated with a low dose of Treprostinil sodium. Dose was escalated to an approximate target dose of 3 ng/kg/min after the first 12 weeks and kept stable for another 12 weeks.
  Due to the predefined infusion rate setting schedule an interim dose of up to 6 ng/kg/min could be reached for few days at the end of the phases 1,2 and 3.
  This depended on the patient's exact weight and is caused by the limited infusion rate setting possibility of the infusion pump.
  Interventions: Drug: Treprostinil sodium

INTERVENTIONS:
Drug: Treprostinil sodium

SUMMARY:
The primary purpose of this study is to determine the effect on six-minute walking test (6MWT) distance after 24 weeks treatment with subcutaneous (SC) Treprostinil Sodium in patients with Severe (inoperable) Chronic Thromboembolic Pulmonary Hypertension.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension (CTEPH) is characterized by non-resolving organized thromboembolic obstructing the pulmonary vascular bed. These thrombi are resistant to thrombolytic therapy and chronic plasmatic anticoagulation. An increase in pulmonary vascular resistance (PVR), right ventricular overload, and eventually right ventricular failure ensue.

The treatment of choice for CTEPH is pulmonary endarterectomy (PEA), providing a potential cure for the disease. However, about 50 % of patients are not candidates for surgery, mainly because of distal location of thromboemboli. Despite recent advances in the treatment of pulmonary arterial hypertension (PAH), medical treatments have not been recommended for inoperable CTEPH, because of the concept that a predominantly major vessel obstructive arteriopathy would not be suitable for vasodilators. Furthermore, a major drawback of i.v. prostacyclin therapy is the need for a permanent central venous access that increases the risk of infection (0.22-0.68 per patient per year), thrombosis and new major vessel thromboembolism.

ELIGIBILITY:
1. Subject must be competent to understand the information given in the written informed consent and from the investigator and must sign and date the informed consent prior to any study mandated procedure.
2. Subject must be at least 18 years of age and can be of any ethnical origin
3. Women of child bearing potential must be surgically sterile or postmenopausal (amenorrhea for at least 12 months) or using an acceptable form of contraception. Reliable contraception is defined as a method which results in a low failure rate, i.e., less than 1% per year when used correctly such as, implants, injectables, oral contraceptive medications, sexual abstinence, or a vasectomised partner.
4. Subject must have a current diagnosis of CTEPH, as defined by the following criteria:

   * A test result of perfusion scintigraphy and pulmonary angiography and/or multislice CT not older than 6 months, consistent with the diagnosis CTEPH. In case of recurrent PH after PEA, test results from before the surgery are acceptable if a typical specimen was harvested during PEA substantiating the diagnosis of CTEPH.
   * A right heart catheterization, not older than 6 months, consistent with the diagnosis CTEPH but specifically with a mean pulmonary artery pressure (PAPm) of > 25 mmHg, and a PVR of > 300 dyn.s.cm-5
   * At least three months of effective anticoagulation therapy (without improvement / to exclude subacute pulmonary emboli)
5. Subject must have CTEPH classified as severe, as defined by the following criteria:

   * An un-encouraged 6MWT distance of between 150 and 400 meters
   * Classification in the WHO/New York Heart Association (NYHA) functional class III or IV
6. The subject must not be suitable to undergo a PEA and is therefore defined as non-operable, due to at least one of the following reasons:

   * Clot is not accessible
   * Discrepancy between severity of PH and morphologic lesion
   * Subject is not a good surgical candidate for other reasons:

   PVR > 1500 dynes.s.cm-5 Age Comorbidity No functional lung parenchyma
   * Unsuccessful PEA in the past with residual/recurrent CTEPH
   * No consent for PEA given by subject
7. Subject must be willing and able to follow all study procedures

Exclusion:

1. Subject with any form of pulmonary arterial hypertension or any disease known to cause PAH (WHO Group I)
2. Subjects with a total lung capacity (TLC) of < 70% predicted or a forced expiratory volume/forced vital capacity (FEV1/FVC < 50%)
3. Subject who received any prostanoids, within the 30 days before screening or be scheduled to receive prostanoids during the course of the study
4. Subject with a new type of chronic therapy (a different category of vasodilator or diuretic) for PAH added within the last month, except anticoagulants
5. Subject with an increased risk for hemorrhage or stroke or with a major cardiovascular event during the past 6 months.
6. Unstable subjects for any reason (according to the investigators discretion)
7. Subject who received any investigational medication within 30 days prior to the screening visit of this study or be scheduled to receive another investigational drug during the course of this study
8. Subject with a known intolerance to any drug relevant for this trial, especially to Treprostinil sodium or prostanoids
9. Subject with a history or suspicion of non compliance
10. Subject who has any musculoskeletal disease or any other disease that would limit ambulation
11. Subject with other cardiovascular, liver, renal, hematologic, gastrointestinal immunologic, endocrine, metabolic, or central nervous system disease that, in the opinion of the investigator, may adversely affect the safety of the subject and /or efficacy of the study drug or limit the lifespan of the subject
12. Female who is considering pregnancy or who is pregnant and/or lactating
13. Subject who is an investigator or any other team member involved directly or indirectly in the conduct of the clinical study.
14. Subject who is an inmate of a psychiatric ward, prison or is suspected not to be able to give consent of his free will

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-03; Primary Completion 2016-11 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Lang, MD, Principal Investigator — Medical University Vienna
Locations (6):
- Austria (2):
  - Krankenhaus der Elisabethinen, Linz
  - Medical University of Vienna AKH - Division Cardiology, Vienna
- II. interní klinika Všeobecná fakultní nemocnice, Prague, Czechia
- Medical University Carl Gustav Carus Medizinische Klinik und Poliklinik I Medizinische Fakultät der Technischen Universität Dresden, Dresden, Germany
- Poland (2):
  - Department of Cardiac and Vascular Diseases Centre for Rare Cardiovascular Diseases John Paul II Hospital, Krakow
  - NZOZ Europejskie Centrum Zdrowia Otwock, Otwock

REFERENCES:
- [Background] Lang IM, Marsh JJ, Olman MA, Moser KM, Loskutoff DJ, Schleef RR. Expression of type 1 plasminogen activator inhibitor in chronic pulmonary thromboemboli. Circulation. 1994 Jun;89(6):2715-21. doi: 10.1161/01.cir.89.6.2715. PMID 8205686
- [Background] Klepetko W, Mayer E, Sandoval J, Trulock EP, Vachiery JL, Dartevelle P, Pepke-Zaba J, Jamieson SW, Lang I, Corris P. Interventional and surgical modalities of treatment for pulmonary arterial hypertension. J Am Coll Cardiol. 2004 Jun 16;43(12 Suppl S):73S-80S. doi: 10.1016/j.jacc.2004.02.039. PMID 15194182
- [Background] McLaughlin VV, Presberg KW, Doyle RL, Abman SH, McCrory DC, Fortin T, Ahearn G; American College of Chest Physicians. Prognosis of pulmonary arterial hypertension: ACCP evidence-based clinical practice guidelines. Chest. 2004 Jul;126(1 Suppl):78S-92S. doi: 10.1378/chest.126.1_suppl.78S. PMID 15249497
- [Background] Kuhn KP, Byrne DW, Arbogast PG, Doyle TP, Loyd JE, Robbins IM. Outcome in 91 consecutive patients with pulmonary arterial hypertension receiving epoprostenol. Am J Respir Crit Care Med. 2003 Feb 15;167(4):580-6. doi: 10.1164/rccm.200204-333OC. Epub 2002 Nov 21. PMID 12446266
- [Derived] Sadushi-Kolici R, Jansa P, Kopec G, Torbicki A, Skoro-Sajer N, Campean IA, Halank M, Simkova I, Karlocai K, Steringer-Mascherbauer R, Samarzija M, Salobir B, Klepetko W, Lindner J, Lang IM. Subcutaneous treprostinil for the treatment of severe non-operable chronic thromboembolic pulmonary hypertension (CTREPH): a double-blind, phase 3, randomised controlled trial. Lancet Respir Med. 2019 Mar;7(3):239-248. doi: 10.1016/S2213-2600(18)30367-9. Epub 2018 Nov 23. PMID 30477763

RESULTS

PARTICIPANT FLOW:
Groups:
- Treprostinil Sodium High Dose (~30ng/kg/Min): Treprostinil sodium was administered subcutaneously via an ambulatory infusion pump with continuous flow rate. Patients were uptitrated to a target dose of approx. 30ng/kg/min within the first 12 weeks and were kept on stable dose for the remaining 12 weeks study duration.
- Treprostinil Sodium Low Dose (~3ng/kg/Min): Treprostinil sodium was administered subcutaneously via an ambulatory infusion pump with continuous flow rate. Patients were uptitrated to a target dose of approx. 3ng/kg/min within the first 12 weeks and were kept on stable dose for the remaining 12 weeks study duration.
Period: Overall Study
Arm/Group | Treprostinil Sodium High Dose (~30ng/kg/Min) | Treprostinil Sodium Low Dose (~3ng/kg/Min)
Started | 53 | 52
Completed | 45 | 46
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- High Dose: Treprostinil sodium high dose
- Low Dose: Treprostinil sodium low dose
- Total: Total of all reporting groups
Arm/Group | High Dose | Low Dose | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 15 | 26 | 41
  >=65 years | 38 | 25 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.06 (11.16) | 60.58 (14.59) | 64.35 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 30 | 49
  Male | 34 | 22 | 56
Region of Enrollment [Number; unit: participants]
  Austria | 28 | 26 | 54
  Czechia | 17 | 17 | 34
  Poland | 8 | 8 | 16
  Germany | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in 6-minute Walk Test Distance After 24 Weeks
Description: To determine the effect of subcutaneous Treprostinil sodium on 6-minute walk test distance after 24 weeks in patients with severe non-operable chronic thromboembolic pulmonary hypertension severe (inoperable) Chronic Thromboembolic Pulmonary Hypertension
  Time frame of the 6-minute walk test: The 6-minute walk test was conducted at the following visits:
  * baseline (day 1)
  * Visit 6 (day 168)
  In case of missing values, Last-Observation-Carried-Forward imputation method was used. In such cases values documented at Visit 4 (day84) were used.
Time Frame: Baseline and 24 weeks
Population: All randomized subjects who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: m
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 53 | 52
m | 45.43 (71.29) | 3.83 (56.21)
Statistical Analysis 1: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.002, ANCOVA
Statistical Analysis 2: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.0003, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Participants With Clinical Worsening
Description: Clinical worsening defined as a decrease of 6-minute walk test distance of more than 20% from baseline due to Chronic Thromboembolic Pulmonary Hypertension, decrease of New York Heart Association functional class, hospitalization with the requirement for additional Pulmonary Hypertension specific treatment and/or death due to worsening Chronic Thromboembolic Pulmonary Hypertension.
  Clinical Worsening was assessed after 12 weeks and 24 weeks, participants experiencing clinical worsening at any time-point are reported.
Time Frame: 12 weeks and 24 weeks
Population: All randomized subjects who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 53 | 52
Participants | 7 | 12
Statistical Analysis 1: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.605, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Effect on Maximal Borg Score During 6-minutes Walk Test
Description: The Borg scale was used for rating of dyspnea during 6-minutes walk test. The scale is defined from 0 to > 10 (upper bound) (0 = NOTHING AT ALL; 0.5 = VERY VERY SLIGHT (just noticeable); 1 = VERY SLIGHT; 2 = SLIGHT; 3 = MODERATE; 4 = SOMEWHAT SEVERE; 5 = SEVERE; 6-9 = VERY SEVERE; 10 = VERY VERY SEVERE (almost maximum); >10 MAXIMUM).
  As can be seen with the scale, the higher scale values represent a worse outcome.
  As no imputation rule applied only full-data sets were evaluated. Complete data sets were available for 48 patients randomized to high dose group and 48 patients in low dose group.
Time Frame: Baseline and 24 weeks
Population: For this endpoint no imputation role was applied. For 48 patients of the high dose group, as well as for the low dose group, baseline data and also 24 week data are available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 48 | 48
units on a scale | -0.44 (2.21) | -0.13 (2.43)
Statistical Analysis 1: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.307, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in WHO/NYHA (World Health Organization - New York Heart Association) Functional Class
Description: Class I - Patients with pulmonary hypertension but without resulting limitation of physical activity. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain or near syncope.
  Class II - Patients with pulmonary hypertension resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain or near syncope.
  Class III - Patients with pulmonary hypertension resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes undue dyspnea or fatigue, chest pain or near syncope
  Class IV - Patients with pulmonary hypertension in the inability to carry out any physical activity without symptoms. These patients manifest signs of right heart failure. Dyspnea and/or fatigue may even be present at rest. Discomfort is increased by any physical activity.
Time Frame: Baseline and 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 53 | 52
Participants
  Improved | 27 | 9
  No change | 22 | 36
  Worse | 2 | 3
  Not done | 2 | 4
Statistical Analysis 1: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.0019, Chi-squared

5. Secondary Outcome: Effect on Quality of Life by the MINNESOTA Questionnaire
Description: This questionnaire is composed of 21 questions relating to limitations in lifestyle associated with Heart Failure. Respondents use a 5-point scale that ranges from 0 (none) to 5 (too much), with a score of 0 representing no limitation and a score of 5 representing maximum limitation. The change in individual score sum was evaluated and is displayed in the results, with a possible range of 0-105. Higher values indicate more limitations in Quality of Life.
  As no imputation rule applied only full-data sets were evaluated. Complete data sets were available for 50 patients randomized to high dose group and 46 patients in low dose group.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 50 | 46
units on a scale | -6.36 (22.9) | -4.63 (19.34)
Statistical Analysis 1: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.557, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Effect on N-terminal Pro-BNP Levels
Description: baseline values, assessment after 12 and 24 weeks
  As no imputation rule applied only full-data sets were evaluated. Complete data sets were available for 46 patients randomized to high dose group and 46 patients in low dose group.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: percentage change to baseline
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 46 | 46
percentage change to baseline | 0.84 (63.32) | 41.68 (104.2)
Statistical Analysis 1: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.032, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Effect on Hemodynamic Parameter (PVR - Pulmonary Vascular Resistance)
Description: baseline values, assessment after 24 weeks
  As no imputation rule applied only full-data sets were evaluated. Complete data sets were available for 48 patients randomized to high dose group and 47 patients in low dose group.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: dyn.s.cm^-5
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 48 | 47
dyn.s.cm^-5 | -214.23 (324.28) | 72.96 (284.95)
Statistical Analysis 1: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.00001, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Effect on Hemodynamic Parameter (CI - Cardiac Index)
Description: as for outcome 7
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: L/min/m2
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 48 | 47
L/min/m2 | 0.42 (0.9) | -0.16 (0.54)
Statistical Analysis 1: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.000003, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Effect on Hemodynamic Parameter (CO - Cardiac Output)
Description: as for outcome 7
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 48 | 47
L/min | 0.63 (1.47) | -0.22 (1.06)
Statistical Analysis 1: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.00008, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Effect on Hemodynamic Parameter (mPAP - Mean Pulmonary Arterial Pressure)
Description: baseline values, assessment after 24 weeks
  As no imputation rule applied only full-data sets were evaluated. Complete data sets were available for 47 patients randomized to high dose group and 47 patients in low dose group.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 47 | 47
mmHg | -3.36 (8.04) | -0.4 (6.87)
Statistical Analysis 1: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Effect on Hemodynamic Parameter (mRap - Mean Right Atrial Pressure)
Description: as for outcome 7
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 48 | 47
mmHg | 0.65 (5.08) | 2.87 (6.82)
Statistical Analysis 1: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.227, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Effect on Signs & Symptoms of the CTEPH
Description: baseline values, assessment after 24 weeks
Time Frame: Baseline and 24 weeks
Measure: Number; unit: participants
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 53 | 52
participants
  Ascites : Baseline | 2 | 3
  Ascites : Week 24 | 1 | 3
  Nausea/Vomiting : Baseline | 4 | 9
  Nausea/Vomiting : Week 24 | 5 | 9
  Chest pain : Baseline | 13 | 11
  Chest pain : Week 24 | 8 | 3
  Orthopnoea : Baseline | 9 | 9
  Orthopnoea : Week 24 | 3 | 5
  Dizziness : Baseline | 25 | 21
  Dizziness : Week 24 | 11 | 10
  Palpitations : Baseline | 19 | 18
  Palpitations : Week 24 | 9 | 11
  Dyspnoea at rest : Baseline | 7 | 10
  Dyspnoea at rest : Week 24 | 3 | 10
  Paroxysmal nocturnal dyspnoea : Baseline | 7 | 1
  Paroxysmal nocturnal dyspnoea : Week 24 | 4 | 3
  Dyspnoea on exertion : Baseline | 53 | 51
  Dyspnoea on exertion : Week 24 | 46 | 43
  Syncope : Baseline | 3 | 6
  Syncope : Week 24 | 1 | 2
  Fatigue : Baseline | 33 | 37
  Fatigue : Week 24 | 26 | 27
  Thirst : Baseline | 12 | 21
  Thirst : Week 24 | 12 | 13

ADVERSE EVENTS:
Arm/Group | High Dose | Low Dose
All-Cause Mortality (participants affected / at risk) | 2/53 | 1/52
Serious Adverse Events (participants affected / at risk) | 9/53 | 10/52
Other Adverse Events (participants affected / at risk) | 53/53 | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=53) | Low Dose (N=52)
Cardiac failure (Cardiac disorders) | 2 | 1
Dyspnea (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 6 | 1
Syncope (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Incarcerated hernia (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Accute kidney injury (Renal and urinary disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Worsening of pulmonary hypertension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=53) | Low Dose (N=52)
Oedema peripheral (Cardiac disorders) | 7 | 10
Diarrhoea (Gastrointestinal disorders) | 33 | 12
Nausea (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 3 | 3
Decreased appetite (General disorders) | 7 | 0
Flushing (General disorders) | 4 | 4
Infusion site reactions (General disorders) | 25 | 24 — Infusion site reactions include inf. site abscess, inf. site erythema, inf. site haemorrhage, inf. site infection, inf. site inflammation, inf. site irritation, inf. site pruritus, inf. site rash, inf. site reaction, inf. site swelling
Infusion site pain (General disorders) | 39 | 42
Nasopharyngitis (Infections and infestations) | 4 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain in extremities (Musculoskeletal and connective tissue disorders) | 11 | 1
Headache (Nervous system disorders) | 12 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Epistaxis (Vascular disorders) | 1 | 3
Worsening of Pulmonary Hypertension (Vascular disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No